CLINICAL TRIAL: NCT00884559
Title: Brief Leadership Instructions Improve Cardiopulmonary Resuscitation in a High Fidelity Simulation: a Randomised Controlled Trial
Brief Title: Leadership Instructions Improve Cardiopulmonary Resuscitation in a High Fidelity Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ekbb_SH_103
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Cardiopulmonary Resuscitations
Keywords: Leadership; Team building; Resuscitation
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Technical (Active Comparator): Technical Instructions
  Interventions: Other: instruction
- Leadership (Experimental): Leadership-Instructions
  Interventions: Other: instruction

INTERVENTIONS:
Other: instruction — Debriefing

SUMMARY:
Whether teaching leadership with a short debriefing has a positive influence on the performance of cardiopulmonary resuscitation remains largely unknown. The investigators will assess the sustained efficacy of a short leadership debriefing compared to a technical debriefing in a high fidelity simulated cardiopulmonary resuscitation.

DETAILED DESCRIPTION:
Context:

Whether the performance of cardiopulmonary resuscitation can be positively influenced by teaching leadership with a short debriefing remains largely unknown

Objective:

To test the hypothesis that (1) leadership instruction are effective and (2) improved leadership results in better performance in a high fidelity simulated cardiopulmonary resuscitation.

Design:

Prospective, randomized-controlled superiority trial

Setting:

Simulator Center of the University Hospital Basel in Switzerland

Patients or Other Participants:

237 volunteer medical students in teams of 3

Intervention:

During a baseline visit, the medical students participate in a video-taped simulated witnessed cardiac arrest. Participants are randomized to receive thereafter a short video-assisted debriefing focusing either on correct positions of arms and shoulders (technical debriefing) or on leadership and communication to enhance team coordination (leadership debriefing). A follow-up simulation is conducted after 4 months. Leadership utterances, technical skills and the resuscitation performance of the teams are compared based on videotapes coded by two independent researchers.

Main Outcome Measures:

The primary outcomes for this study are the amount of hands-on time in the first 180 seconds after the onset of the cardiac arrest and the time elapsed until cardiopulmonary resuscitation was started. Secondary endpoints are the effectiveness of the technical and leadership instructions, respectively.

ELIGIBILITY:
Inclusion Criteria:

* volunteer medical students

Exclusion Criteria:

* no informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 237 (Actual)
Dates: Start 2005-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Hands-on time in the first 180 seconds after the onset of the cardiac arrest and the time elapsed until cardiopulmonary resuscitation is started. | 180 sec after start of CPR

SECONDARY OUTCOMES:
The effectiveness of the technical and leadership instructions | 180 sec after starting CPR

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Hunziker, MD, Principal Investigator — University Hospital, Basel, Switzerland; Stephan Marsch, Prof, Study Chair — Intensive Care unit, University Hospital Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland